CLINICAL TRIAL: NCT00445172
Title: A Long-Term Study in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E0302-J081-762
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2017-08

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis; Motor Neurons; Muscular Atrophy
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Muscular Atrophy | interventions — mecobalamin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E0302 (mecobalamin)

INTERVENTIONS:
Drug: E0302 (mecobalamin) — Intramuscular injection, mecobalamin twice a week.

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of long-term E0302 administration in patients with Amyotrophic Lateral Sclerosis (ALS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have completed Phase II/III study of E0302 (E0302-J081-761, hereafter referred to as Study 761) except for those patients who discontinued the treatment of Study 761. Completed patients are defined as those who completed the treatment period of Study 761, those on 24-hour use of non-invasive positive pressure ventilation (NIPPV), or those who eventually resulted in the use of NIPPV.
2. Patients who are able to submit written informed consent. If patients are duly capable of study consent but are unable to sign (or affix a seal) by themselves due to aggravation of disease condition, written informed consent can be obtained from a legally authorized representative who can sign on behalf of the patients after confirming the patients' agreement to study participation.

Exclusion Criteria:

1. Patients with cognitive impairment.
2. Pregnant women or women who may have a possibility of becoming pregnant.
3. Patients or their partners who are not willing to use reliable contraception.
4. Patients with severe disease in the renal, cardiovascular, hematological, or hepatic system (severe disease will be judged referring to "Ministry of Health, Labor and Welfare (MHLW) Drug Safety Dept. Notification No. 80, Drug Safety Classification Criteria for Severity of Adverse Drug Reaction by Medicinal Products, Grade 3." However, an event due to the primary disease will be precluded).
5. Patients with malignant tumor.
6. Patients who participated in another clinical study after the completion of Study 761.
7. Patients with present illness or history of drug allergy or severe allergic disease (anaphylactic shock).
8. Patients who are judged to be ineligible for study entry by the investigator or subinvestigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a Measure of safety | Every 3 months

SECONDARY OUTCOMES:
Survival rate | Every 3 months
Functional rating scale | Every 3 months
Percent-predicted forced vital capacity (%FVC.) | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kazunori Saeki, Study Director — Neuroscience Clinical Development Section. JAC PCU. Eisai Co., Ltd.
Locations (42):
- Japan (42):
  - Nagoya, Aichi-ken
  - Aomori, Aomori
  - Chiba, Chiba
  - Touon-shi, Ehime
  - Fukuoka, Fukuoka
  - Kitakyushi-shi, Fukuoka
  - Fukushima, Fukushima
  - Maebashi, Gunma
  - Higashihiroshima-shi, Hiroshima
  - Miyoshi-shi, Hiroshima
  - Otake-shi, Hiroshima
  - Sapporo, Hokkaido
  - Kanazawa, Ishikawa-ken
  - Ichinoseki-shi, Iwate
  - Sagamihara-shi, Kanagawa
  - Yokohama, Kanagawa
  - Nangoku-shi, Kochi
  - Kyoto, Kyoto
  - Tsu, Mie-ken
  - Sendai, Miyagi
  - Watari-gun, Miyagi
  - Nagano, Nagano
  - Higashisonogi-gun, Nagasaki
  - Kashiwazaki-shi, Niigata
  - Niigata, Niigata
  - Tsukubo-gun, Okayama-ken
  - Ginowan-shi, Okinawa
  - Toyonaka-shi, Osaka
  - Hasuda-shi, Saitama
  - Saitama-shi, Saitama
  - Hamamatsu, Shizuoka
  - Shizuoka, Shizuoka
  - Shimotsuke-shi, Tochigi
  - Tokushima, Tokushima
  - Yoshinogawa-shi, Tokushima
  - Bunkyo-ku, Tokyo
  - Kodaira-shi, Tokyo
  - Ōta-ku, Tokyo
  - Wakayama, Wakayama
  - Yonezawa-shi, Yamagata
  - Shimonoseki-shi, Yamaguchi
  - Yanai-shi, Yamaguchi